CLINICAL TRIAL: NCT07256548
Title: Comparative Evaluation of Machine Learning Algorithms for Predicting Spinal Anesthesia Termination Time
Brief Title: Machine Learning for Predicting Spinal Anesthesia Duration
Status: Recruiting | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Principal Investigator, Sıddık Varolgunes, MD, Kocaeli City Hospital
Other Study IDs: KSH_SVG_1
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Spinal Anesthesia; Machine Learning; Knee Arthroplasty, Total; Spinal Anesthesia Duration; Postoperative Care; Postoperative Acute Pain
Keywords: spinal anesthesia; machine learning; Knee arthroplasty; spinal anesthesia duration; Acute postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Spinal; Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Knee Arthroplasty Group: The group of patients who will undergo knee replacement surgery under spinal anesthesia
  Interventions: Procedure: Spinal Anesthesia (bupivacaine)

INTERVENTIONS:
Procedure: Spinal Anesthesia (bupivacaine) — Before being placed on the operating table, the patient is positioned comfortably and prepared for the procedure. Standardized monitoring is initiated, including five-lead electrocardiography (ECG), non-invasive blood pressure (NIBP), and pulse oximetry (SpO₂). Baseline measurements of heart rate, systolic and diastolic blood pressure, mean arterial pressure (MAP), and oxygen saturation are recorded. An 18- or 20-gauge intravenous line is inserted, and an appropriate crystalloid preload is administered. After ensuring aseptic conditions, the patient is positioned in the sitting posture, and spinal puncture is performed at the L3-L4 or L4-L5 intervertebral space using a 25 Gauge Whitacre needle. Following free flow of cerebrospinal fluid, 0.5% hyperbaric bupivacaine (10-15 mg) is slowly injected. The completion of the injection is

SUMMARY:
Spinal anesthesia provides significant advantages over general anesthesia in knee arthroplasty, including reduced blood loss, faster recovery, and fewer complications. However, predicting its duration is critical for patient safety and effective postoperative management. This study evaluates the usability of machine learning (ML) algorithms to predict the termination time of spinal anesthesia and the patient's readiness for mobilization. Using demographic, surgical, and anesthetic variables, ML models were trained to estimate anesthesia duration. Accurate predictions may improve intraoperative planning, optimize postoperative care, and enhance patient outcomes. Integrating ML-based predictive systems into anesthesia practice can contribute to safer, more efficient, and personalized perioperative management.

DETAILED DESCRIPTION:
Abstract

Spinal anesthesia offers several advantages over general anesthesia in total knee arthroplasty, including reduced intraoperative blood loss, less postoperative pain, faster recovery, and shorter hospital stays. It also minimizes anesthesia-related complications and facilitates early mobilization, making it a preferred technique for many orthopedic procedures. However, predicting the exact duration of spinal anesthesia remains challenging and is clinically significant for ensuring patient safety, optimizing postoperative pain control, and preventing anesthesia-related complications.

Accurate estimation of anesthesia duration allows for more effective surgical planning, timely analgesia administration, and improved patient satisfaction. Unexpectedly prolonged anesthesia may increase the risk of adverse effects, whereas premature termination can result in inadequate pain management.

Machine learning (ML) technologies offer promising tools for predicting clinical outcomes in anesthesia practice by analyzing complex, multidimensional datasets. Previous research has demonstrated the potential of ML algorithms to predict perioperative events such as hypotension, blood transfusion requirements, and postoperative complications.

In this study, the usability and effectiveness of ML models in predicting the time of termination of spinal anesthesia and the patient's readiness for mobilization were investigated. By incorporating multiple clinical variables-such as patient demographics, anesthetic drug dosages, and surgical factors-our model aims to provide accurate, data-driven predictions. These predictive insights can support anesthesiologists in tailoring perioperative management, reducing complication risks, and improving overall patient outcomes. Ultimately, integrating ML-based prediction systems into anesthesia practice may enhance the safety, efficiency, and personalization of perioperative care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled to undergo total knee arthroplasty between November 2025 and March 2026 at the Kocaeli City Hospital Operating Theaters.
2. Patients who have provided written informed consent to participate in the study.
3. Patients whose surgery is planned under spinal anesthesia.
4. Patients for whom complete clinical data can be obtained during the study period.
5. Adults aged 18 years or older, classified as American Society of Anesthesiologist's (ASA) Physical Status I or II.

Exclusion Criteria:

1. Patients who were converted to general anesthesia during surgery or initially operated under general anesthesia.
2. Patients who required postoperative intensive care unit (ICU) admission following anesthesia.
3. Patients who developed surgical complications and for whom postoperative mobilization could not be planned.
4. Patients with cognitive impairment preventing them from completing pain assessment scales in the postoperative period.
5. Patients with neuropathic pain, multiple sclerosis, or other neuromotor disorders will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients undergoing elective total knee arthroplasty (TKA) under spinal anesthesia at Kocaeli City Hospital Operating Theaters between November 2025 and March 2026.
  All participants will receive spinal anesthesia using 0.5% hyperbaric bupivacaine, and intraoperative monitoring will be conducted in accordance with institutional anesthesia standards. The study population represents a homogeneous surgical group in which spinal anesthesia is routinely applied, allowing for standardized anesthesia protocols and reliable measurement of anesthesia duration.
  Eligible patients will be classified as ASA Physical Status I or II and aged 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Predictive performance of machine learning | From the end of intrathecal injection (T₀) to complete motor recovery (T_end), expected within 6 hours post-injection.
  The primary outcome of this study is the predictive performance of machine learning (ML) algorithms in estimating the duration of spinal anesthesia (in minutes) based on preoperative and intraoperative variables.
  in: R² (Coefficient of Determination). Dimensionless (no unit)

SECONDARY OUTCOMES:
spinal anesthesia termination time | From the end of intrathecal injection (T₀) to complete motor recovery (T_end), expected within 6 hours post-injection.
  It is the period of time from the moment of completion of spinal anesthesia until the complete resolution of motor blockade in the patient's lower extremities.
Visual Analogue Scale | From the end of intrathecal injection (T₀) to complete motor recovery (T_end), expected within 6 hours post-injection.
  A tool used to help a person rate the intensity of certain sensations and feelings, such as pain. The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. It may be used to help choose the right dose of pain medicine.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Yüksek, MD, Study Director — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, İzmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bellini V, Russo M, Domenichetti T, Panizzi M, Allai S, Bignami EG. Artificial Intelligence in Operating Room Management. J Med Syst. 2024 Feb 14;48(1):19. doi: 10.1007/s10916-024-02038-2. PMID 38353755
- [Background] Cao Y, Wang Y, Liu H, Wu L. Artificial intelligence revolutionizing anesthesia management: advances and prospects in intelligent anesthesia technology. Front Med (Lausanne). 2025 Aug 6;12:1571725. doi: 10.3389/fmed.2025.1571725. eCollection 2025. PMID 40842529
- [Background] Magdic Turkovic T, Sabo G, Babic S, Sostaric S. SPINAL ANESTHESIA IN DAY SURGERY - EARLY EXPERIENCES. Acta Clin Croat. 2022 Sep;61(Suppl 2):160-164. doi: 10.20471/acc.2022.61.s2.22. PMID 36824644
- [Background] Boublik J, Gupta R, Bhar S, Atchabahian A. Prilocaine spinal anesthesia for ambulatory surgery: A review of the available studies. Anaesth Crit Care Pain Med. 2016 Dec;35(6):417-421. doi: 10.1016/j.accpm.2016.03.005. Epub 2016 Jun 21. PMID 27352633
- [Background] Schubert AK, Wiesmann T, Wulf H, Dinges HC. Spinal anesthesia in ambulatory surgery. Best Pract Res Clin Anaesthesiol. 2023 Jun;37(2):109-121. doi: 10.1016/j.bpa.2023.04.002. Epub 2023 Apr 15. PMID 37321760